CLINICAL TRIAL: NCT05672745
Title: An Open-label Pilot Study to Learn How the Phenotypical Characteristics of Woebot Users Are Related to Clinical Outcomes
Brief Title: How Phenotypical Characteristics of Woebot Users Are Related to Clinical Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woebot Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: W-LIFE-001
Record Dates: First submitted 2022-12-13; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: To Understand the Characteristics of Digital Mental Health Intervention Users as They Relate to Mental Health Outcomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WB-LIFE (Experimental)
  Interventions: Device: WB-LIFE

INTERVENTIONS:
Device: WB-LIFE — WB-LIFE is a mobile application program grounded in validated psychotherapies (including cognitive behavioral therapy, interpersonal, and dialectical behavioral therapy), that enlists the relational agent Woebot to guide users in managing their mood. The user experience is driven by artificial intelligence and centers around mood tracking, evidence-based tools, and goal-oriented, tailored conversations.

SUMMARY:
The goal of this observational study is to understand the characteristics of Woebot users as they relate to clinical outcomes.

The objectives it aims to address are:

1. To assess Woebot usage patterns, satisfaction ratings, self-efficacy, stress, resilience, work productivity and activity impairment, alexthymia, and bond over time based on demographic, clinical baseline levels, and attitudinal characteristics
2. Among users who present with clinical levels of anxiety or depression, to assess the contribution of demographic characteristics, attitudinal characteristics, and patterns of engagement on clinical outcomes of interest over time
3. To collect and explore attitudinal characteristics of Woebot users regarding their experiences with mental health care and perceived value of digital tools for emotional support
4. Explore meaningful subgroups of Woebot users based on demographic and attitudinal characteristics, clinical outcomes, and patterns of engagement

Participants who meet study eligibility requirements will be:

* invited to engage with the Woebot Life program for 8 weeks
* complete survey assessments at day 3, week 4 (mid-intervention), and week 8 (end of intervention)

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* US resident
* English literacy
* Availability to complete survey assessments
* Ownership or regular access to a smartphone with WiFi and sufficient data access for the duration of the study.

Exclusion Criteria:

* Current suicidal ideation with a plan or intent or a suicide attempt within the past 12 months
* A reported lifetime diagnosis of a psychotic disorder (including schizophrenia or schizoaffective disorder) or bipolar disorder
* Previous use of the Woebot application

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-07-23 (Actual); Study Completion 2022-07-23 (Actual)

PRIMARY OUTCOMES:
App engagement metrics | Baseline to Post-intervention at Week 8
  Data tracking mobile application use, including conversational interactions with Woebot and patterns of engagement over time, will be collected throughout the duration of treatment (8-weeks).
Client Satisfaction Questionnaire (CSQ-8) | Post-intervention at Week 8
  An 8-item measure used to assess client's satisfaction with treatment.Total scores range from 8-32, with high scores indicating greater satisfaction with the treatment.
Working Alliance Inventory (WAI) | Change from Day 3 to Mid-Intervention at Week 4; change from Day 3 to Post-intervention at Week 8; change from Mid-Intervention at Week 4 to Post-intervention at Week 8
  Measure of working alliance. A measure of therapeutic alliance that assesses three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. Total scores range from 12-60, with higher scores indicating greater alliance. The present study utilized the validated 12-item Short-Revised version (WAI-SR) with minor changes to language, replacing "therapist" with "Woebot".
Mental Health Self-Efficacy Scale (MHSES) | Change from Baseline to Mid-Intervention at Week 4; change from Baseline to Post-intervention at Week 8; change from Mid-Intervention at Week 4 to Post-intervention at Week 8
  Six items assess confidence in managing stress, depression, and anxiety, and are scored on a 10 point Likert scale (from 1, not at all confident to 10, very confident). Ratings across the 6 items are summed for an overall measure of MHSES (range 10 to 60), with higher scores indicating more self-efficacy. This measure is included as a way to capture an individual's confidence that they can successfully manage their mental health concerns.
Patient-Reported Outcomes Measurement Information System Global Health (PROMIS) | Change from Baseline to Mid-Intervention at Week 4; change from Baseline to Post-intervention at Week 8; change from Mid-Intervention at Week 4 to Post-intervention at Week 8
  Ten items used to assess five core domains of health (physical function, pain, fatigue, emotional distress, and social). Total scores range from 5-50, where greater scores represent the best health and functioning.
Patient Health Questionnaire | Change from Baseline to Mid-Intervention at Week 4; change from Baseline to Post-intervention at Week 8; change from Mid-Intervention at Week 4 to Post-intervention at Week 8
  Measure of depression. An 8-item self-report questionnaire where total scores range from 0 to 24, with higher scores indicating greater levels of depression
Generalized Anxiety Disorder Questionnaire | Change from Baseline to Mid-Intervention at Week 4; change from Baseline to Post-intervention at Week 8; change from Mid-Intervention at Week 4 to Post-intervention at Week 8
  Measure of anxiety. A 7-item brief self-report questionnaire, where total score range is between 0-21, with higher scores indicate greater levels of anxiety.
Brief Resilience Questionnaire (BRS) | Change from Baseline to Mid-Intervention at Week 4; change from Baseline to Post-intervention at Week 8; change from Mid-Intervention at Week 4 to Post-intervention at Week 8
  The BRS is a measure used to assess a person's ability to bounce back or recover after experiencing a stressor. Total scores range from 1 (low resilience) to 5 (high resilience).
Perceived Stress Scale (PSS) | Change from Baseline to Mid-Intervention at Week 4; change from Baseline to Post-intervention at Week 8; change from Mid-Intervention at Week 4 to Post-intervention at Week 8
  The PSS is a 10-item tool to assess individual levels of stress in the past month. Total scores range from 0 (no stress) to 40 (very high levels of stress).
Toronto Alexithymia Scale (TAS) | Change from Baseline to Mid-Intervention at Week 4; change from Baseline to Post-intervention at Week 8; change from Mid-Intervention at Week 4 to Post-intervention at Week 8
  The TAS-20 is an instrument that measures alexithymia, or difficulty with identifying and describing emotions and focusing attention externally. Total scores range from 20-100, with with low levels of alexithymia indicative of high levels of emotional self-awareness and vice versa.
Work Productivity and Activity Impairment (WPAI) | Change from Baseline to Mid-Intervention at Week 4; change from Baseline to Post-intervention at Week 8; change from Mid-Intervention at Week 4 to Post-intervention at Week 8
  The WPAI measures presenteeism, absenteeism, work productivity loss for the currently employed, and activity impairment.
  WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity
Burnout | Change from Baseline to Mid-Intervention at Week 4; change from Baseline to Post-intervention at Week 8; change from Mid-Intervention at Week 4 to Post-intervention at Week 8
  Single-item question to measure burnout on a scale from 1-5, where 5 is feeling completely burned out to the point change is needed.

SECONDARY OUTCOMES:
Perceived Barriers to Care (PBC) | Day 3 of Intervention
  The PBC is a 30-item assesses perceived barriers to access mental health care on a scale of 1= not at all to 5 = impossible, including Stigma, Lack of motivation, Emotional concerns, Negative evaluations of therapy, Misfit of therapy to needs, Time constraints, Participation restriction, Availability of Services, and Cost.
Woebot Attitudinal Survey (WAS) | Post-intervention at Week 8
  The 9-item survey was designed to assess the user's perceptions of their Woebot experience - perceptions of skills learned, emotional challenges addressed, relational quality (comprehension of information, relevance of suggestions offered, perceptions of support, lack of judgment), applications of Woebot suggestions in daily life, and perceptions about the session duration and length of engagement with Woebot app needed for Woebot to work effectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Woebot Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiauzzi E, Williams A, Mariano TY, Pajarito S, Robinson A, Kirvin-Quamme A, Forman-Hoffman V. Demographic and clinical characteristics associated with anxiety and depressive symptom outcomes in users of a digital mental health intervention incorporating a relational agent. BMC Psychiatry. 2024 Jan 30;24(1):79. doi: 10.1186/s12888-024-05532-6. PMID 38291369
- [Derived] Hoffman V, Flom M, Mariano TY, Chiauzzi E, Williams A, Kirvin-Quamme A, Pajarito S, Durden E, Perski O. User Engagement Clusters of an 8-Week Digital Mental Health Intervention Guided by a Relational Agent (Woebot): Exploratory Study. J Med Internet Res. 2023 Oct 13;25:e47198. doi: 10.2196/47198. PMID 37831490
- [Derived] Forman-Hoffman VL, Pirner MC, Flom M, Kirvin-Quamme A, Durden E, Kissinger JA, Robinson A. Engagement, Satisfaction, and Mental Health Outcomes Across Different Residential Subgroup Users of a Digital Mental Health Relational Agent: Exploratory Single-Arm Study. JMIR Form Res. 2023 Sep 27;7:e46473. doi: 10.2196/46473. PMID 37756047